CLINICAL TRIAL: NCT01090544
Title: Transnasal Insufflation for Patients With COPD GOLD IV and Hypercapnia
Brief Title: Transnasal Insufflation (TNI) and Chronic Obstructive Pulmonary Disease
Acronym: TNICOPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Helios Klinik Ambrock (Other)
Responsible Party: Georg Nilius MD, Helios Klinik Hagen Ambrock
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Helios TNI 2010
Record Dates: First submitted 2010-03-19; First posted 2010-03-22 (Estimated); Last update posted 2010-09-30 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; TNI; PaCO2
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Nasal Insufflation — Breathing therapy
  Other Names: TNI 20 oxy

SUMMARY:
The purpose of this study is to determine wether transnasal insufflation as an alternate form of breathing support for COPD patients will lead to improvement of their medical condition.

DETAILED DESCRIPTION:
Chronic obstructive pulmonary disease (COPD) is a slowly proceeding lung disease which basic pathophysiologic mechanisms are only partly understood so far and which is difficult to access with a pharmacological or sundry approach besides smoking cessation. Average life expectancy is clearly limited especially in advanced stages with respiratory insufficiency . Based on different smaller surveys long-term oxygen treatment is classified to be the routine in COPD treatment when patients develop hypoxemia.

The primary application of non-invasive ventilation Routine is the treatment for COPD patients with acute respiratory decompensation and developing hypoxemia and respiratory acidosis, because it reduces the acute mortality as various prospective randomized studies showed.

On the other side there are no distinct informations and data about the initiation of a nocturnal positive pressure breathing therapy when chronic hypercapnia appear in progression of COPD.

Nocturnal positive pressure therapy appliqued with a mask can be assumed to be the routine treatment for neuromuscular and restrictive thorax diseases, because nocturnal ventilation results in a distinct increase of life expectancy.

In contrast data about positive pressure therapy at COPD are inconsistent and initiation of nocturnal breathing therapy is practised in many places, but is scientifically not confirmed yet.

It is known from various other studies with other patient collectives with nocturnal positive pressure therapy, like patients with obstructive sleep apnoea syndrome, that only 50 to 70% of those patients are using their therapy constantly. Daily practice shows that patients with chronic hypercapnia based on COPD are even harder to accustom oneself to a nocturnal breathing therapy than patients with restrictive lung diseases or patients with obstructive sleep apnoea syndrome.

Reasons for that are not known, but maybe the significant lung distension or increased appearance of depressive or anxiety disorders of COPD patients are responsible for that.

Perhaps patients do not feel a subjective improvement of their medical condition and don't accept a tight closing mask at nights.

As a result an alternate form of breathing support would be desirable.

ELIGIBILITY:
Inclusion Criteria:

* COPD GOLD IV
* PCO2 > 50 mmHg
* competent patients
* stable respiratory situation

Exclusion Criteria:

* serious acute diseases
* hypercapnic decompensation pH < 7,30

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
partial pressure of carbon dioxide (PaCO2) decrease | 3 hours
  PaCO2 is measured before and after applying TNI, and a PaCO2 decrease is supposed to be assessed.

SECONDARY OUTCOMES:
Breathing Frequency | 3 hours
  Breathing Frequency is supposed to decrease under TNI treatment

CONTACTS AND LOCATIONS:
Overall Officials: Georg Nilius, MD, Principal Investigator — Helios Klinik Hagen Ambrock
Locations (1):
- Helios Klinik Hagen Ambrock, Hagen, North Rhine-Westphalia, Germany